CLINICAL TRIAL: NCT01161433
Title: Implementing Evidence-based Quality Improvement Strategies to Improve Asthma Care for Children
Brief Title: A Practical Model to Transform Childhood Asthma Care - Spirometry Training in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: James W. Stout/Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 32583-E/B; HHSA290200600022, Task order 2 (Other Grant/Funding Number: Agency for Healthcare Research and Quality)
Record Dates: First submitted 2010-06-15; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Asthma
Keywords: Asthma; Spirometry; Pediatric; Primary Health Care; Education, Distance
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Virtually delivered spirometry quality improvement program
  Interventions: Behavioral: Virtually delivered spirometry quality improvement program
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Virtually delivered spirometry quality improvement program — Sites in the intervention arm receive the virtually delivered QI program.
  The program includes:
  1. Spirometry Fundamentals™ CD-ROM, a computer-based CD-ROM training program that teaches primary care providers and their staff techniques required to perform high-quality spirometry tests, and proper interpretation of spirometric data;
  2. Case-based, interactive webinars; and
  3. an Internet-based spirometry quality feedback reporting system.
  Arms: Intervention

SUMMARY:
Spirometry is a recommended component of asthma diagnosis and treatment in the primary care setting, however, few primary care providers report routine use of spirometry in the provision of care for their asthma patients. Even when spirometry is used to aid in asthma severity classification, primary care providers have a high rate of failing to meet the quality goals for testing established by the American Thoracic Society.

The goal of this study is to evaluate the effectiveness of a virtually delivered quality improvement (QI) program. The program is designed to train primary care providers and their medical staff in the use of spirometry to improve pediatric primary care management for children with asthma.

DETAILED DESCRIPTION:
A cluster randomized trial with matched practice pairs. All practices receive a spirometer and standard vendor training. Those randomized to the intervention group receive a 7-month QI program, which includes:

1. Spirometry Fundamentals™ CD-ROM;
2. Case-based, interactive webinars; and
3. an Internet-based spirometry quality feedback reporting system.

ELIGIBILITY:
Inclusion Criteria:

* Internet access on a computer running Windows XP SP2
* Access to a computer with Windows 2000 /Mac OS 10 or higher
* Practices must match another enrolled practice on the following parameters.

  1. Number of providers in practice (same number +/- 1 provider)
  2. Location - both practices must either be urban or rural
  3. % of patients eligible for Medicaid (same percentage +/- 15%)
  4. Practice type (school-based clinic, Federally Qualified Health Center, private practice, hospital- or university-based clinic)
  5. Geographic distance (minimum of 10 miles away from matched pair practice)

Exclusion Criteria:

* Lack of Internet access on a computer running Windows XP SP2
* Lack of access to a computer with Windows 2000 /Mac OS 10 or higher
* Practices that were unable to be matched to another similar practice

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Spirometry test quality | Seven months
  Percentage of acceptable quality spirometry tests as determined by standards set by the American Thoracic Society.

SECONDARY OUTCOMES:
Presence of asthma care plan | Seven months
  To assess whether exposure to the virtually delivered quality improvement (QI) program increases the frequency with which written asthma action plans are completed.
Asthma severity documentation | Seven months
  To assess whether exposure to the virtually delivered quality improvement (QI) program increases the frequency with which asthma severity is appropriately documented.
Appropriate prescription of controller therapy | Seven months
  To assess whether exposure to the virtually delivered quality improvement (QI) program increases the frequency with which appropriate controller therapy is prescribed.
Frequency of office-based spirometry | Seven months
  To test whether exposure to the virtually delivered quality improvement (QI) program increases the frequency with which office-based spirometry is used in the management of children with asthma.

CONTACTS AND LOCATIONS:
Overall Officials: James W Stout, MD, MPH, Principal Investigator — University of Washington; Rita Mangione-Smith, MD, MPH, Principal Investigator — University of Washington/Seattle Children's Hospital
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: Spirometry 360 Training Program — http://depts.washington.edu/imtr/spiro360/